CLINICAL TRIAL: NCT02387944
Title: "Point-Of-Care" Evaluation of Hemostasis in Children With Congenital Heart Disease
Brief Title: Bedside Evaluation of Coagulation in Children With Congenital Heart Disease
Acronym: POCHEMO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, David Longchamp, PICU consultant, MD, Centre Hospitalier Universitaire Vaudois
Other Study IDs: 468/14
Record Dates: First submitted 2015-03-05; First posted 2015-03-13 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Congenital Heart Defect; Blood Coagulation Disorder
Keywords: Children; Cyanotic congenital heart defect; Cardiopulmonary Bypass; Thromboelastometry; Platelet Function Tests
MeSH Terms: conditions — Heart Defects, Congenital; Blood Coagulation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cardiopulmonary bypass: Children with congenital heart defect undergoing surgery on cardiopulmonary bypass
- cardiac catheterism: Children with congenital heart defect undergoing cardiac catheterism

SUMMARY:
The purpose of this study is to assess coagulation and platelet function in children with congenital heart disease, measured with a bedside device (thromboelastometry and impedance aggregometry).

The investigators also aim to determine if this device detect post-cardiopulmonary bypass clotting derangements and may help to manage bleeding in this population.

DETAILED DESCRIPTION:
Hemostasis, a main concern during and after any surgical procedure, is traditionally monitored by the following laboratory tests: activated Partial Thrombin Time (aPTT), prothrombin time (PT), fibrinogen, platelets count. They neither provide a reliable estimate of the risk of bleeding, nor allow determining useful interventions.

New investigations of hemostasis are now used and validated during and after surgery: Rotational Thromboelastometry (ROTEM®) and impedance aggregometry. This is a quick bedside functional analysis of the patient's clotting. Children who undergo surgery under cardiopulmonary bypass (CPB) are particularly at risk of bleeding and this population hasn't been studied with large cohort yet.

Hypothesis: Hemostasis in children with CHD, especially when cyanotic, is intrinsically abnormal. The corrective surgery on CPB induces further hemostatic disorders which can be identified by the ROTEM platelet®.

The aim of the study is to evaluate the hemostatic function of the child with congenital heart disease using a Point-Of-Care (platelet-ROTEM ®) system, before surgery and after alterations induced by cardiopulmonary bypass (CPB).

This is a single center, observational, prospective study. Expected duration: 2 years. The investigators plan to include 200 patients with CHD, 100 patients undergoing surgery with CPB and 100 patients with congenital heart disease requiring cardiac catheterization. Recruitment will be conducted by the Division of Paediatric Cardiology.

Inclusion criteria include an age of 0-16 years and a diagnosis of congenital heart disease requiring surgery with CPB or cardiac catheterization. Patients with known dyscrasia or treated with antiaggregant within 10 days/oral anticoagulants within 48h before surgery/catheterization.

ROTEM platelet® test will be performed before surgery/catheterization. Patients undergoing surgery will have a second test within 30 minutes after the end of cardiopulmonary bypass. All patients will benefit from the usual cares.

ELIGIBILITY:
Inclusion Criteria:

* children between 0 and 16 years, born with a congenital heart disease requiring either cardiac catheterization or surgery with cardiopulmonary bypass
* parental and/or patient consent

Exclusion Criteria:

* known hemostatic disorder
* known platelet function disorder
* antiaggregation treatment <10 days before blood sampling
* oral anticoagulation <2 days before blood sampling
* intravenous heparin <6 hours before blood sampling
* patient and parents unable to consent

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with congenital heart defect
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-03; Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Hemostasis measured by thromboelastometry and impedance aggregometry | Single measurement, during general anesthesia, immediately before procedure, when arterial line available
Hemostasis measured by thromboelastometry and impedance aggregometry in cyanotic children | Single measurement, during general anesthesia, immediately before procedure, when arterial line available

SECONDARY OUTCOMES:
Thromboelastometry and impedance aggregometry changes after cardiopulmonary bypass (CPB) | maximum 3 measurements, during surgery and up to 6 hours after end of CBP
Thromboelastometry and impedance aggregometry changes in children with significant bleeding after CPB | Single measurement, during general anesthesia, immediately before procedure, when arterial line available

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Di Bernardo, MD, Principal Investigator — CHUV
Locations (1):
- PICU, Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Longchamp D, Perez MH, Natterer J, Amiet V, Ferry T, Boegli Y, Mauron S, Dolci M, Plaza Wuthrich S, Di Bernardo S. Point-of-care hemostasis in children with congenital heart disease, the POCHEMO study: baseline reference values of thromboelastometry and impedance aggregometry. Blood Coagul Fibrinolysis. 2019 Jul;30(5):199-204. doi: 10.1097/MBC.0000000000000818. PMID 31157681